CLINICAL TRIAL: NCT03587545
Title: Study of Probiotic Potential of Nasopharyngeal Lactobacillus Strains in the Upper Respiratory Tract After Nasal Spray Application
Brief Title: Study of Probiotic Potential of Lactobacillus Strains in the Upper Respiratory Tract After Nasal Spray Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité, UZA, Principal Investigator, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: B300201835709
Record Dates: First submitted 2018-06-27; First posted 2018-07-16 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers; Chronic Rhinosinusitis (Diagnosis); Probiotics; Sprays; Nasal Disease
MeSH Terms: conditions — Disease; Nose Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Healthy probiotic group LGG (Experimental): Daily intake by healthy volunteers of 2 dosages of LGG spray during 2 weeks. Probiotic nasal spray.
  Interventions: Other: Probiotic nasal spray
- Healthy probiotic group LAMBR2 (Experimental): Daily intake by healthy volunteers of 2 dosages of LAMBR2 spray during 2 weeks. Probiotic nasal spray.
  Interventions: Other: Probiotic nasal spray
- Healthy placebo group (Placebo Comparator): Daily intake by healthy volunteers of 2 dosages of placebo spray during 2 weeks.
  Placebo nasal spray.
  Interventions: Other: Placebo nasal spray
- CRS probiotic group LGG (Experimental): Daily intake by CRS patients of 2 dosages of LGG spray during 2 weeks. Probiotic nasal spray.
  Interventions: Other: Probiotic nasal spray
- CRS probiotic group LAMBR2 (Experimental): Daily intake by CRS patients of 2 dosages of LAMBR2 spray during 2 weeks. Probiotic nasal spray.
  Interventions: Other: Probiotic nasal spray
- CRS placebo group (Placebo Comparator): Daily intake by CRS patients of 2 dosages of placebo spray during 2 weeks. Placebo nasal spray.
  Interventions: Other: Placebo nasal spray

INTERVENTIONS:
Other: Probiotic nasal spray — Total daily nasal administration of 2*10^8 CFU of probiotic bacteria delivered via 2 servings.
  Arms: CRS probiotic group LAMBR2; CRS probiotic group LGG; Healthy probiotic group LAMBR2; Healthy probiotic group LGG
Other: Placebo nasal spray — Two servings of nasal administration of placebo nasal spray (not containing probiotic bacteria)
  Arms: CRS placebo group; Healthy placebo group

SUMMARY:
Probiotics are defined as "live micro-organisms that, when administered in adequate amounts, confer a health benefit to the host" (Hill et al, 2014). These microbes are generally applied in the gastrointestinal tract via fermented food products or capsules. In previous research, the investigators isolated bacterial strains with potential probiotic properties for the upper respiratory tract based on in vitro laboratory tests, in vivo mice experiments and genome sequencing.

In this study, the investigators want to deliver the Proof-of-Concept that the most promising isolated strain, Lactobacillus casei AMBR2 (LAMBR2) and the well-documented probiotic strain Lactobacillus rhamnosus GG (LGG) also have interesting properties in humans, i.e. that these strains are able to -temporarily- persist in the upper respiratory tract of healthy volunteers and CRS patients after daily nasal application via a nasal spray for 2 weeks. In addition, the investigators aim to explore whether the application of these strains has an impact on the nasopharyngeal microbiome via 16S rRNA amplicon sequencing and dedicated qPCR analysis.

Therefore, bacterial DNA from nasal swabs will be isolated via commercially available DNA extraction kits, followed by Illumina MiSeq sequencing in order to identify the bacterial species present in these samples. Furthermore, the concentration of the Lactobacillus and specific pathogens will be monitored via qPCR.

ELIGIBILITY:
Inclusion Criteria:

* CRS patient group: CRS diagnosed

Exclusion Criteria:

* no patients with trisomy 21
* no pregnant women
* no breastfeeding women
* no acute or chronic airway infections (except for CRS patients in CRS patient group)
* no cancer
* no autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Nasal persistence of lactobacilli | 3 years
  After DNA extraction of the biological samples, the relative and absolute concentration of the administered probiotics will be monitored via microbiome analysis and qPCR. This will give information about the capacity of the probiotics to colonize the nasopharynx.

SECONDARY OUTCOMES:
Microbiome differences | 3 years
  After Illumina MiSeq sequencing, bio-informatic tools will be used to cluster bacteria into amplicon sequence variants (ASVs). Based on these ASVs, the investigators will compare the composition of the bacteria in the sampled niches and compare this composition between patient with and without intake of probiotics. The investigators will specifically screen for ASVs that are over- or underrepresented in both populations. Furthermore, special attention will go to screen for the typical nasopharyngeal pathogens such as Staphylococcus aureus, Streptococcus pneumoniae, Haemophilus influenzae, Moraxella catarrhalis... and also to beneficial microbes such as lactic acid bacteria.
Therapeutic potential: chronic rhinosinusitis | 3 years
  Chronic rhinosinusitis symptoms will be evaluated before and after administration of the nasal spray. Participants should rate the complaints linked to CRS from 'not present' to 'serious'.
Therapeutic potential: nasal hyperreactivity | 3 years
  Nasal hyperreactivity symptoms will be evaluated before and after administration of the nasal spray.
Therapeutic potential: SNOT-22 score | 3 years
  The investigators will investigate whether the nasal intake of probiotics has an effect on the quality of life of CRS patients. Patients should rate general nasopharyngeal complaints from 0 to 5 where 0 means that there is no complaint and 5 means that there are serious complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lebeer, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://procureproject.be/en/